CLINICAL TRIAL: NCT00645554
Title: A Bioequivalent Study to Compare Galantamine Oral Solution With Marketed Galantamine Capsule After Single Oral Administration of 10 mg.
Brief Title: A Single Dose, Cross-over Bioequivence Study Comparing Galantamine IR (Immediate Release) Table and Galantmine OS (Oral Solution) in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Xian-Janssen Pharmaceutical Ltd. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR002848
Record Dates: First submitted 2008-03-24; First posted 2008-03-27 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2010-03

CONDITIONS: Pharmacokinetics
Keywords: Galantamine oral solution; Galantamine tablet; Bioequivalence
MeSH Terms: interventions — Galantamine

INTERVENTIONS:
Drug: Galantamine oral solution

SUMMARY:
The purpose of this open-label, single dose, two-treatment, two-period, cross-over study is to evaluate the pharmacokinetic profile and tolerability of galantamine oral solution and galantamine tablet.

DETAILED DESCRIPTION:
This is an open-label, single dose, two-treatment, two-period, cross-over study to evaluate the pharmacokinetic profile and tolerability of galantamine oral solution and galantamine tablet. All patients are healthy male patients who are 18-45 years old with BWI (Body Weight Index) between 18-28 kg/m2. All patients must sign informed consent before being enrolled. 24 patients were randomized in the study. The duration of study is 9 days. All patients must stay at site unit for 12 hours after single oral administration otherwise patients could stay home but must return to site at specific date and time. The day before dosing day (baseline), patients were randomized to one of the two groups to be administered either 4mg galantamine oral solution (1ml) or galantamine tablet (1 tablet). After 7-day washout period, patients were crossed over to receive the other formulation. Pharmacokinetic observation will last to 32 hours after dosing. Plasma were collected at immediately before dosing and 0.25, 0.5, 0.75, 1.5, 2, 3, 4, 6, 8, 12, 24 and 32 hours after dosing to determine plasma concentration of galantamine. Safety and tolerance evaluation will last until Day 9. Safety evaluation include adverse events, vital signs, physical examination, electrocardiogram and laboratory tests. On study Day 1, patients will take either 4mg galantamine oral solution (1ml) or 4mg galantamine tablet (1 tablet). After 7-day washout period, on Day 8, patients will cross over to take the other formulation, the dosage and administration are the same.

ELIGIBILITY:
Inclusion Criteria:

* All patients must meet the following criteria: body weight index is between 18-28 kg/m2
* Patients are deemed healthy based on physical examination, medical history, vital signs, electrocardiogram and results of clinical laboratory tests
* All patients must be able to read and understand the contents of informed consent that must be signed prior to any trial-specific procedures are done.

Exclusion Criteria:

* Patients meeting one or more of the following criteria cannot be included in the study: the patient uses disallowed medicine, which is any prescribed medication within the last 2 weeks or OTC drugs within the last week prior to dosing (or at least 5 half lives for any drug ingested). Patients who have taken any non-prescribed systemic or topical medication may still be entered into the study, if, in the opinion of the investigator, the medication will not interfere with the study procedures or compromise safety
* The subject has history of alcohol or drug abuse
* Patient has been treated with an investigational drug within 30 days prior to screening
* Patient has a know hypersensitivity to galantamine or has a history of severe drug allergy or hypersensitivity
* Patient has any serious illness such as liver or renal insufficiency, cardiovascular, pulmonary, gastrointestinal, endocrine, neurological, metabolic and other chronic disturbance
* Patient has donated blood within 60 days prior to dosing
* Patient is a moderate or severe smoker who smokes more than 3 cigarettes, or ex-smokers who has ceased smoking for at least 3 months prior to dosing
* Patient, in the opinion of the investigator, is unlikely to comply with the clinical study protocol or is unsuitable for any other reason

Ages: 18 Years to 48 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
It is estimated that the plasma maximal concentration of galantamine (Cmax=31.53mg×L-1) after single oral administration can be reached in Chinese young volunteers at the peak time of 1.66 hours. The half life is 7.06 hours.

SECONDARY OUTCOMES:
The relative bioavialibility of galantamine oral solution (4mg) indicated by AUC0-t and AUC0-inf are 105.6%±18.5% and 106.2%±19.5% respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Xian-Janssen Pharmaceutical Ltd. Clinical Trial, Study Director — Xian-Janssen Pharmaceutical Ltd.

REFERENCES:
- See also: A bioequivalent study of galantamine oral solution comparing with galantamine tablet in healthy Chinese male subjects — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=1076&filename=CR002848_CSR.pdf